CLINICAL TRIAL: NCT03269461
Title: Serial OCT Evaluation of Tissue Coverage in Patients Submitted to Inspiron Drug Eluting Stent Implantation
Acronym: REPAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REPAIR
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease
Keywords: stent, DES, INSPIRON, OCT, tissue repair
MeSH Terms: conditions — Coronary Artery Disease; Dysequilibrium syndrome; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 days evaluation (Experimental): Angiography and Optical Coherence Tomography evaluations
  Interventions: Device: Angiography and Optical Coherence Tomography evaluations
- 2 months evaluation (Experimental): Angiography and Optical Coherence Tomography evaluations
  Interventions: Device: Angiography and Optical Coherence Tomography evaluations
- 3 months evaluation (Experimental): Angiography and Optical Coherence Tomography evaluations
  Interventions: Device: Angiography and Optical Coherence Tomography evaluations

INTERVENTIONS:
Device: Angiography and Optical Coherence Tomography evaluations — coronary stent implantation followed by Angiography and Optical Coherence Tomography evaluations

SUMMARY:
Prospective, multicentric, single-arm study to evaluate fast and effective tissue repair in patients undergone percutaneous coronary intervention with drug eluting stent Inspiron.

DETAILED DESCRIPTION:
The first 20 patients enrolled will be evaluated by angiography and Optical Coherence Tomography 3 months after stent implantation. The following 20 patients will be evaluated by the same methods 2 months after the implantation and the last 20 patients after 30 days.

All patients will be clinically followed at 30 days, 6 months, 1 and 2 years after index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 80years;
* Symptomatic CAD or documented myocardial ischemic disease;
* Up to 2 de novo lesions on native coronary arteries;
* Lesion length ≤ 29mm;
* Reference vessel diameter between ≥2.5 and ≤ 3.5 mm;
* Stenose at target lesion ≥ 70% and ≤ 99%.

Exclusion Criteria:

* STEMI within the last 72 hours pre-procedure;
* renal insufficiency;
* Left Main stenosis > 50%;
* Ostial lesions;
* Bifurcation lesions with side branch ≥2mm;
* More than one lesion > 50% at the target vessel;
* Left Ejection Fraction less than 30%;
* Previous (less than 6 months) PCI at the target vessel.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Tissue Coverage | 3 months
  Change in the tissue coverage percentage measured by OCT

SECONDARY OUTCOMES:
in-stent late lumen loss | 3 months
  in-stent late lumen loss
Stent Thrombosis | 2 years
  Stent Thrombosis Rates
Target Vessel Failure | 2 years
  Target Vessel Failure (Death, MI and new revascularization)

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Hospital Evangélico do Espírito Santo, Vila Velha, Espírito Santo
  - Hospital do Coração Anis Rassi, Goiânia, Goiás
  - Paraná Medical Research Center, Maringá, Paraná
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No